CLINICAL TRIAL: NCT00487877
Title: Measurements of Skin Physiological Parameters as Mean of Metabolic Assessment
Acronym: TEMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TASMC-06-NV-380-CTIL
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2006-12

CONDITIONS: Hungry-Satiation Situation
Keywords: metabolism, temperature changing, skin, heart rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SenseWear Pro3 Armband
Device: i-button DS2191 H

SUMMARY:
To investigate the relationship between hungry-satiation situation including meal time and metabolism, skin temerature changing, simpathetic & para-simpathetic response To investigate the relashionship between hungry-satiation situation including meal time and heart rate

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. BMI: 22-30 Kg / m2

Exclusion Criteria:

1. Any unbalanced chronic disease
2. Any infection disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof., Principal Investigator — unaffiliation; Nachum Vaisman, Prof., Principal Investigator
Locations (1):
- The Unit of clinical Nutrition, Tel Aviv, Israel